CLINICAL TRIAL: NCT06971172
Title: EFFECT OF LOW LEVEL LASER THERAPY ON ORAL PIMPHIGUS VULGARIS
Brief Title: Low-level Laser Therapy on Oral Pemphigus Vulgaris Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, University doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: low energy laser in pemphigus
Record Dates: First submitted 2024-12-08; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Pemphigus Vulgaris
MeSH Terms: conditions — Pemphigus | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low energy laser plus medical treatment (Experimental): Device
  Interventions: Device: Low energy diode Laser
- Medical treatment (Active Comparator): Medical treatment
  Interventions: Drug: Medication

INTERVENTIONS:
Device: Low energy diode Laser — Diode Laser
  Arms: Low energy laser plus medical treatment
Drug: Medication — pulse steriod therapy and immunosuppressive drugs
  Arms: Medical treatment

SUMMARY:
To assess the therapeutic efficacy of low level laser therapy on oral pemphigus vulgaris patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oral pemphigus vulgaris

Exclusion Criteria:

* other causes of oral ulcers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
wound margins in millimeters | 1 month
  Measurement